CLINICAL TRIAL: NCT03025126
Title: Human Empowerment Aging and Disability (HEAD): New Technologies for Neurorehabilitation
Acronym: HEAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Centro Riabilitativo Villa Beretta (Unknown); Fondazione Opera S Camillo (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FdG_HEAD_01
Record Dates: First submitted 2017-01-12; First posted 2017-01-19 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-01

CONDITIONS: Rehabilitation; Technology; Telerehabilitation; Nervous System Diseases
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- HEAD Rehabilitation (Experimental): rehabilitation with IT multimedial devices
  Interventions: Other: Multimedial Rehabilitation
- Usual care program (Active Comparator): usual care program
  Interventions: Other: Usual care program

INTERVENTIONS:
Other: Multimedial Rehabilitation
  Arms: HEAD Rehabilitation
Other: Usual care program — Usual care at home program according to healthcare professional's advice
  Arms: Usual care program

SUMMARY:
Congenital or acquired neurological disorders could lead to consistent motor and cognitive disabilities. The continuity and persistency of a tailored home rehabilitation protocol after recovery is crucial to prevent disease aggravation or relapses. The integration of a web-based new technology in home rehabilitation programme can constitute a functional low cost resource by offering patients off-line (and on-line) monitoring and by proposing new motivating ways of rehabilitation through high tech tools such as serious games.

ELIGIBILITY:
Inclusion Criteria:

* age range 18-85
* Parkinson Disease (PD - mild to moderate) in stable treatment for at least 3 months
* Multiple Sclerosis (MS) without relapses in the last 3 months (EDSS ≤ 6)
* post stroke ( ≥ 6 months after the acute event)

Exclusion Criteria:

* Mini Mental State Examination < 20
* limited range of motion
* severe pain
* severe deficit of visual acuity or auditory perception or communication and severe dysmetry

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03; Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life assessed on the short-form 12-item Health Survey (SF-12) questionnaire | change from baseline after 4 months and after 7 months
Global cognitive state assessed on MONTREAL COGNITIVE ASSESSMENT (MOCA) | change from baseline after 4 months and after 7 months
Endurance assessed on two-minute walking test (2MWT) | change from baseline after 4 months and after 7 months
Positive and negative affective state assessed on Positive and Negative Affect Scale (PANAS) | change from baseline after 4 months and after 7 months

SECONDARY OUTCOMES:
Static balance and fall risk assessed on Berg Balance Scale (BBS) | change from baseline after 4 months and after 7 months
Finger dexterity assessed on 9-Hole Peg Test (9HPT) | change from baseline after 4 months and after 7 months
Unilateral gross manual dexterity assessed on Box and Blocks Test (BBT) | change from baseline after 4 months and after 7 months
Walking speed assessed on 10-Meter Walking Test (10MWT) | change from baseline after 4 months and after 7 months
Strength in upper and lower extremities assessed on Motricity Index (MI) | change from baseline after 4 months and after 7 months
Attention and concentration assessed on Attention and Concentration test | change from baseline after 4 months and after 7 months
Memory abilities assessed on Rivermead Behavioural Memory Test - 3 (RBMT3) | change from baseline after 4 months and after 7 months
Caregiver Need assessed on Caregiver Need Assessment (CNA) questionnaire | change from baseline after 4 months and after 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Franco Molteni, MD, Principal Investigator — Valduce Hospital
Locations (3):
- Italy (3):
  - Ospedale Valduce, Lecco, LC
  - Presidio Sanitario S Camillo, Torino, TO
  - Fondazione Don Carlo Gnocchi ONLUS, Milan

REFERENCES:
- [Derived] Jonsdottir J, Baglio F, Gindri P, Isernia S, Castiglioni C, Gramigna C, Palumbo G, Pagliari C, Di Tella S, Perini G, Bowman T, Salza M, Molteni F. Virtual Reality for Motor and Cognitive Rehabilitation From Clinic to Home: A Pilot Feasibility and Efficacy Study for Persons With Chronic Stroke. Front Neurol. 2021 Apr 7;12:601131. doi: 10.3389/fneur.2021.601131. eCollection 2021. PMID 33897579